CLINICAL TRIAL: NCT02890407
Title: Genetics of Aortic Stenosis: From Family Forms to the Common Forms
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/09/61
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The association study will compare the allele frequencies of polymorphisms of a single nucleotide (SNP) in the population of individuals with aortic stenosis compared to a control population.

Patients will be included only if they are suffering from a typical form of tight and surgical tricuspid aortic stenosis. Patients will therefore only included if they are suffering from aortic stenosis, the surface is less than 1 cm² and if histological analysis or failing intraoperative findings of the surgeon showed a tricuspid aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria has reached:

   * That patients are operated or not, they can be considered as having a degenerative aortic stenosis, patients will be diagnosed with aortic stenosis (aortic area <1 cm) without obvious cause found.
2. criteria not met

   * Strictly normal aortic valve by ultrasound in an over 65-year-old patient.
   * All patients do not fit into the above two categories are considered as having an unknown phenotype and will not be used in binding assays. In particular, the presence of an aortic sclerosis or even moderate aortic regurgitation can be considered as potentially incipient form of aortic stenosis, patients with this type of anomaly will not be scanned during family analyzes.

Exclusion Criteria:

* Patients who did not sign the consent
* Non degenerative aortic stenosis or for which another cause could be found.

Among the most commonly found causes are:

* Bicuspid aortic valve
* Severe renal impairment
* Severe Hypercholesterolemia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 1. Criteria has reached:
     * That patients are operated or not, they can be considered as having a degenerative aortic stenosis, patients will be diagnosed with aortic stenosis (aortic area <1 cm) without obvious cause found.
  2. criteria not met
     * strictly normal aortic valve by ultrasound in an over 65-year-old patient.
Sampling Method: Probability Sample
Enrollment: 1987 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
identify the genetic factors involved in the occurrence of aortic stenosis | 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CHU de Nantes -, Nantes
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boureau AS, Karakachoff M, Le Scouarnec S, Capoulade R, Cueff C, de Decker L, Senage T, Verhoye JP, Baufreton C, Roussel JC, Dina C, Probst V, Schott JJ, Le Tourneau T. Heritability of aortic valve stenosis and bicuspid enrichment in families with aortic valve stenosis. Int J Cardiol. 2022 Jul 15;359:91-98. doi: 10.1016/j.ijcard.2022.04.022. Epub 2022 Apr 13. PMID 35427703